CLINICAL TRIAL: NCT02150512
Title: Resuscitation Strategies in Septic Shock. A Randomized Controlled Trial of Two Different Fluid Loading Strategies in ICU Patients With Early Septic Shock
Brief Title: Resuscitation Strategies in Septic Shock
Acronym: ReSSeS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medisch Spectrum Twente (Other)
Responsible Party: Principal Investigator, RJ Trof, MD PhD, Medisch Spectrum Twente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ReSSeS-2014
Record Dates: First submitted 2014-05-19; First posted 2014-05-30 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Septic Shock; Critically Ill
Keywords: Septic shock; Critically ill patients; Transpulmonary thermodilution; Fluid resuscitation
MeSH Terms: conditions — Shock, Septic; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transpulmonary thermodilution (TPTD) (Experimental): The intervention group (TPTD guided therapy) follows a fluid resuscitation protocol based on stroke volume variation (SVV) and extravascular lung water (EVLW). Initial trigger for fluid loading when circulatory insufficiency is present will be SVV.
  Interventions: Device: Transpulmonary Thermodilution
- Surviving Sepsis Guidelines (SSG) (Active Comparator): The standard group (SSG guided therapy) follows a fluid resuscitation protocol based on the Surviving Sepsis Campaign recommendations. Initial trigger for fluid loading when circulatory insufficiency is present will be the CVP (target ≥12 mmHg).
  Interventions: Device: Surviving Sepsis Guidelines (SSG)

INTERVENTIONS:
Device: Transpulmonary Thermodilution — Initial trigger for fluid loading when circulatory insufficiency is present will be SVV. If SVV ≤10% in patients on controlled mechanical ventilation with tidal volumes of ≥8 ml/kg, fluid loading will not be performed. If SVV >10% or spontaneous breathing efforts are present, a fluid challenge should be performed. Also if patients are on controlled mechanical ventilation with tidal volumes of ≤7 ml/kg, a fluid challenge should be performed. If fluid responsiveness is present and SVV decreases to ≤10%, further fluid loading should be stopped. If SVV is still >10%, the increase in EVLW will decide whether to continue fluid loading or not; if EVLW is ≥12 mL/kg PBW and EVLW increases upon fluid loading, further fluid loading should be stopped.
  Other Names: PiCCO, Pulsion Medical Systems, Germany
  Arms: Transpulmonary thermodilution (TPTD)
Device: Surviving Sepsis Guidelines (SSG) — Initial trigger for fluid loading when circulatory insufficiency is present will be the CVP (target ≥12 mmHg). If circulatory insufficiency is absent, fluid loading will not be initiated or stopped independently of the actual CVP level.
  Arms: Surviving Sepsis Guidelines (SSG)

SUMMARY:
The purpose of this study, in mechanically ventilated septic shock patients, is to determine whether a fluid loading strategy based on parameters derived from the transpulmonary thermodilution technique may lead to more ventilator free days compared to a fluid loading strategy based on the surviving sepsis guidelines.

DETAILED DESCRIPTION:
Rationale: Fluid loading is an important intervention in patients with severe sepsis and septic shock in order to prevent development of multi organ failure and mortality. The Surviving Sepsis Guidelines recommend during the first 6 hours of resuscitation a central venous pressure (CVP) based fluid loading approach, targeting to 12-15 mmHg in mechanically ventilated patients. CVP however has proven to be a poor indicator for preload and preload dependency, while dynamic parameters as stroke volume variation (SVV) derived from the transpulmonary thermodilution technique (TPTD) are superior. Together with the ability to measure the extravascular lung water (EVLW), the TPTD technique may guide fluid management more accurately and may prevent deleterious fluid overloading.

Objective: The risk of fluid overloading in mechanically ventilated patients with septic shock is less when fluid administration is based on a fluid loading protocol using SVV together with EVLW measurements than applying the Surviving Sepsis Guidelines targeting CVP to 12-15 mmHg, in at least the first 6 hours of resuscitation, translating in more ventilator free days (VFDs) Study design: This is a prospective, randomized, non-blinded, single-center, controlled clinical trial comparing two different fluid resuscitation strategies in patients with septic shock. Patients will be randomized for fluid management based on the Surviving Sepsis Guidelines (SSG) or based transpulmonary thermodilution (TPTD) derived SVV and EVLW in at least the first 6 hours of resuscitation.

Study population: All patients of ≥18 years admitted to the ICU because of septic shock together with the need for mechanical ventilation are eligible for randomization Intervention: During at least the first 6 hours of resuscitation, the standard group (SSG guided therapy) follows a fluid resuscitation protocol based on the Surviving Sepsis Campaign recommendations. Initial trigger for fluid loading when circulatory insufficiency is present will be the CVP (target ≥12 mmHg). The intervention group (TPTD guided therapy) follows a fluid resuscitation protocol based on SVV and EVLW. Initial trigger for fluid loading when circulatory insufficiency is present will be SVV. The study protocol will be applied up to a maximum of 72 hours.

Main study parameters/endpoints: VFDs on day 28. Benefit and risks associated with participation: Since inclusion criteria include a TPTD (5F fiber optic, femoral artery) catheter, the inconvenience as compared to standard treatment is minimal. Current routine hospital policy involves TPTD catheter insertion in most of the patients meeting the inclusion criteria specified above.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Clinical evidence of sepsis (microbiology confirmation, radiological or direct view (pus in biological fluid) or direct surgical view).
3. ≥ 2 SIRS criteria:

   1. Temperature < 36.0°C or > 38.0°C
   2. Heart rate > 90 bpm
   3. Respiratory rate > 20 rpm or PaCO2 < 4.2 kPa or need of mechanical ventilation.
   4. Leukocytes > 12.0 x109/L or < 4.0 x109/L or >10% bands
4. Circulatory shock defined as sustained systemic hypotension (systolic arterial pressure <90 mmHg or MAP <65 mmHg (<75 mmHg in a hypertensive patient) despite a 1,000 ml IV fluid challenge over 30 min (including IV fluids administered pre-ICU) or the need for vasopressor therapy. Hypertensive patients are patients with a history of confirmed hypertension treated with antihypertensive agents.
5. Mechanical ventilation by endotracheal tube (any form)

Exclusion Criteria:

1. Pregnancy
2. Pre-terminal illness with life expectancy <28 days
3. Duration of circulatory shock >6 hours
4. Severe peripheral arterial vascular occlusion disease (Fontaine level III-IV)
5. Inability for femoral artery canulation
6. No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
ventilator free days (VFDs) | 28 days
  VFDs from enrolment to extubation until day 28

SECONDARY OUTCOMES:
duration of circulatory shock (hours) | 72 hours
  Duration of circulatory shock, defined as the amount of consecutive hours on vasopressor therapy

OTHER OUTCOMES:
mortality | 30 days and 90 days
  ICU mortality plus 30-days and 90-days mortality
RIFLE-F score | 5 days
  Evolution of renal function (RIFLE-F score) during the first 5 days after inclusion and use of renal replacement therapy (RRT)
fluid balance | 5 days
  Fluid balances during the first 5 days after inclusion
length of stay in the ICU | 28 days
  Length of stay in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: RJ Trof, MD PhD, Principal Investigator — Medisch Spectrum Twente, department of Intensive Care; A Beishuizen, MD PhD, Study Director — Medisch Spectrum Twente, department of Intensive Care
Locations (1):
- Medisch Spectrum Twente, Enschede, Netherlands